CLINICAL TRIAL: NCT07170930
Title: The Effect of a Training Programme in the Variation of Fitness Parameters, Physiological, Hematological and Biochemical Indicators of Soccer Players During the Preseason Period
Status: Enrolling by invitation | Type: Observational
Sponsor: Emmanouil D. Zacharakis (Other)
Responsible Party: Sponsor-Investigator, Emmanouil D. Zacharakis, PhD, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Other Study IDs: ERC-002/2023
Record Dates: First submitted 2025-07-01; First posted 2025-09-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Athletic Performance; Soccer; Muscle Damage; Inflammation; Exercise Test; Pre-season Training; Exercise Physiology; Physical Fitness; Exercise-induced Inflammation
Keywords: Pre-season training; Match-play exposure; Physiological adaptation; Biochemical markers; Recovery strategies; Training intensity; Physiological stress; Football; Aerobic-anaerobic; Effect; Athletic; Performance adaptation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood (for haematological, endocrine, inflammatory, and muscle damage markers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extended-Play: Participants with higher cumulative friendly match-play exposure during the late pre-season phase.
  Interventions: Other: Friendly Match-Play Exposure: extended vs. limited
- Limited-Play: Participants with lower cumulative friendly match-play exposure during the late pre-season phase.
  Interventions: Other: Friendly Match-Play Exposure: extended vs. limited

INTERVENTIONS:
Other: Friendly Match-Play Exposure: extended vs. limited — This research explores the multidimensional physiological and biochemical responses to differing volumes of friendly match-play (i.e., extended vs. limited) during the late pre-season phase in soccer players.

SUMMARY:
The goal of this study is to investigate the effects of varying friendly match-play exposure during the late pre-season on physiological, biochemical, and performance adaptations in soccer players. It is hypothesized that (i) significant changes will occur across the pre-season in both the extended- and limited-play groups when analysed independently; (ii) distinct group-specific adaptations will emerge by the end of the preparatory period; and (iii) match-play exposure, when analysed across all participants, will be significantly correlated with physiological and performance outcomes at pre-season completion. Players from a randomly selected team will be assessed at three time points: pre-season start, mid-pre-season (MPS), and pre-competition phase (PC). Assessments will include anthropometry, physical performance, and markers of muscle damage, inflammation, hormonal status, and haematology. Based on the total match-play time of 8 friendly games during the late pre-season, players will be retrospectively categorised into extended-play (EP) and limited-play (LP) cohorts.time of 8 friendly games during the late pre-season, players will be retrospectively categorised into extended-play (EP) and limited-play (LP) cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* Aged 18 years or older
* Non-smokers
* Injury-free for the past 6 months
* Medication-free for the past 6 months
* Abstinent from alcohol
* Living at an altitude below 1500 meters
* Committed exclusively to soccer (no participation in other sports)

Exclusion Criteria:

* History of serious injuries (e.g., fractures, ligament tears) within the past 6 months
* Chronic medical conditions such as cardiovascular disease, diabetes, or respiratory disorders
* Current use of performance-enhancing drugs or supplements
* Participation in non-soccer-related sports or activities during the study period

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants are highly active soccer players (i.e., >1000 MET-min·week-¹) and compete at national-level standards.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Body Mass | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Body mass measured at standard anatomical sites using a calibrated scale to track longitudinal changes over the pre-season.
  Unit of Measure: kg
Body Fat | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Body fat percentage measured using skinfold calipers at standard sites to monitor longitudinal changes.
  Unit of Measure: %
Rate of Perceived Exertion (RPE) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Participants rate exertion during standardized training sessions using the Borg Scale (6 = no exertion, 20 = maximal exertion).
  Unit of Measure: Borg 6-20 scale
Glucose | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Fasting blood glucose measured to track metabolic changes over pre-season.
  Unit of Measure: mg/dL
Cholesterol | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Total serum cholesterol measured to assess lipid profile adaptations.
  Unit of Measure: mg/dL
Triglycerides | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum triglycerides measured to monitor metabolic response to training.
  Unit of Measure: mg/dL
SGOT (AST) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum glutamic-oxaloacetic transaminase measured to assess liver/muscle stress.
  Unit of Measure: U/L
SGPT (ALT) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum glutamic-pyruvic transaminase measured to monitor liver/muscle stress.
  Unit of Measure: U/L
Creatine Phosphokinase (CPK) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: CPK measured to detect skeletal muscle damage.
  Unit of Measure: U/L
Myoglobin | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Myoglobin measured as a marker of muscle damage.
  Unit of Measure: ng/mL
Iron | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum iron measured to assess iron status.
  Unit of Measure: µg/dL
Ferritin | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum ferritin measured to monitor iron storage.
  Unit of Measure: ng/mL
C-Reactive Protein (CRP) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: CRP measured as a marker of systemic inflammation.
  Unit of Measure: mg/L
High-sensitivity CRP (hs-CRP) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: hs-CRP measured to detect low-grade inflammation.
  Unit of Measure: mg/L
Interleukin-6 (IL-6) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: IL-6 measured from serum to assess inflammatory response.
  Unit of Measure: pg/mL
Tumor Necrosis Factor-alpha (TNF-α) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: TNF-α measured as a marker of systemic inflammation.
  Unit of Measure: pg/mL
Testosterone | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum testosterone measured to assess hormonal adaptations.
  Unit of Measure: ng/dL
Cortisol | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Serum cortisol measured to monitor stress response.
  Unit of Measure: µg/dL
Testosterone-Cortisol Ratio | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Calculated ratio to estimate anabolic-catabolic balance.
  Unit of Measure: Ratio
Red Blood Cells (RBC) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: RBC count measured from blood to assess oxygen transport capacity.
  Unit of Measure: million cells/µL
Hemoglobin | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Hemoglobin measured to evaluate oxygen-carrying capacity.
  Unit of Measure: g/dL
Hematocrit | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Hematocrit measured as percentage of RBC in blood.
  Unit of Measure: %
White Blood Cells (WBC) | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: WBC count measured to monitor immune function.
  Unit of Measure: cells/µL
Platelets | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Platelet count measured to assess hematological health.
  Unit of Measure: cells/µL
Countermovement Jump Height | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Jump height measured (cm) to assess lower-limb explosive power.
  Unit of Measure: cm
Knee Extensor Power, Dominant Leg | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Measured using isokinetic dynamometer.
  Unit of Measure: Watts
Knee Extensor Power, Non-Dominant Leg | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Measured using isokinetic dynamometer.
  Unit of Measure: Watts
Knee Flexor Power, Dominant Leg | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Measured using isokinetic dynamometer.
  Unit of Measure: Watts
Knee Flexor Power, Non-Dominant Leg | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Measured using isokinetic dynamometer.
  Unit of Measure: Watts
10-m Sprint Time | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Sprint time measured using photocell gates; lower times indicate better performance.
  Unit of Measure: seconds
T-Test Agility | Each measure assessed at Baseline (pre-season start), 4 weeks (mid-pre-season), and 8 weeks (pre-competition phase).
  Description: Participants perform T-test agility course; lower times indicate better agility.
  Unit of Measure: seconds

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education and Sports Science, National and Kapodistrian University of Athens, Athens, Daphni, Greece

IPD SHARING:
Plan to Share IPD: Yes